CLINICAL TRIAL: NCT02692911
Title: Chile Biliary Longitudinal Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999916070; 16-C-N070
Record Dates: First submitted 2016-02-25; First posted 2016-02-26 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2020-06

CONDITIONS: Gallbladder Cancer; Nutritional and Metabolic Diseases
Keywords: Gallbaldder; Cancer; Gallstones; Cholecystectomy; Inflammation
MeSH Terms: conditions — Gallbladder Neoplasms; Nutritional and Metabolic Diseases; Neoplasms; Gallstones; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Women with gallstones: Women aged 50-74 with gallstones

SUMMARY:
Background:

The gallbladder is a small organ below the liver. Gallbladder cancer is a leading cause of cancer death among women in Chile. Chile also has among the highest rates of gallbladder cancer and death in the world. Researchers in a high-risk region of Chile want to find out more about this type of cancer. They especially want to know how inflammation affects the way it develops.

Objective:

To better understand the causes of gallbladder diseases and factors that may be associated with them.

Eligibility:

Women ages 50 74 with gallbladder cancer who are covered by the Chilean national health system.

Other people over age 21 with gallbladder disease.

Healthy adults over age 21.

Design:

Participants may be screened with an ultrasound. They may be asked questions about their health.

Participants will have an ultrasound of the abdomen. This can be done at the study clinic or in the hospital or at home. The ultrasound uses sound waves to take pictures of the gallbladder.

Participants will have a physical exam.

Participants will have their mouths looked at for tooth loss, dentures, and gum redness.

Participants will give a blood sample or saliva sample.

Participants will be asked for access to their medical history. They may be asked to allow researchers to keep any samples taken during gallbladder surgery.

Participants will answer questions about their medical history. This will include illnesses, surgeries, medicine use, and family history. It will also include diet and lifestyle habits, such as places where they have lived and worked.

Some participants will have 3 follow-up visits over 6 years.

...

DETAILED DESCRIPTION:
Gallbladder cancer is a leading cause of cancer death among women in Chile, which has among the highest reported gallbladder cancer incidence and mortality rates in the world. Gallbladder cancer provides a particularly good model for understanding the role of inflammation in carcinogenesis since the major risk factor, gallstones, causes substantial inflammation in the gallbladder. Chile also has a high prevalence of obesity, diabetes, and metabolic syndrome, which are increasingly understood as inflammatory disorders, but the extent to which their carcinogenic effects are mediated through inflammatory pathways is unknown.

While the vast majority of gallbladder cancer cases have gallstones, only a small fraction of gallstone patients ever develop gallbladder cancer. Since there is no way to identify this small proportion at risk, gallstone cases are cholecystectomized, which, given large absolute numbers of individuals with gallstones, results in overtreatment of some and under-treatment of others in a high-risk area like Chile. While cholecystectomy is standard treatment for symptomatic relief, there are more people who need surgery than there are surgeons to perform them, and individuals aged 34-49 are prioritized for treatment, regardless of symptoms. This practice may lead to overtreatment among 34-49-year-olds and under treatment of individuals aged 50 and above since they have to wait longer for surgery. At the same time, about 30% of patients with a biliary colic attack will never have another attack, and cholecystectomy does not always lead to the cessation of symptoms. In addition, cholecystectomy has been associated with an increased risk of other digestive diseases. Thus, cholecystectomy may not be needed in all gallstone patients and may in fact increase the risk of cancer in some. Better predictors of risk are clearly needed.

As with other cancers, dysplasia is an important epidemiologic endpoint as the immediate precursor to cancer since the vast majority of gallbladder cancers develop through a histologic continuum of chronic cholecystitis, pseudopyloric metaplasia, incomplete intestinal metaplasia, dysplasia, and cancer. Thus, our aim is to identify risk factors for gallbladder dysplasia and cancer (GDC) and potential non-invasive risk stratification methods, such as ultrasound characteristics alone or in combination with inflammatory markers and patient characteristics, to better understand the etiology and natural history of GDC and to help inform strategies for GDC prevention.

Together with collaborators at Pontifica Universidad Catolica (PUC), we successfully completed a pilot study in Chile that was previously reviewed and approved by SAG and provided baseline data for the proposed study. Our pilot demonstrated high recruitment rates in the target enrollment area (80%) and high rates of questionnaire completion (100%), blood collection (78% population-based controls), and participant retention (93% of eligible completed a follow-up visit). Information from the pilot was used to optimize procedures for the longitudinal study. We also found that both gallstones and gallbladder cancer were associated with systemic immune alterations, which as we previously demonstrated, reflect inflammatory changes in the gallbladder detectable in bile. The next step is to demonstrate that these markers precede GDC by longitudinally measuring their levels among gallstone patients.

We propose to prospectively assess risk factors and early detection markers for GDC by conducting the Chile Biliary Longitudinal Study (BiLS), a cohort study of 6250 individuals with gallstones from the high- risk southern-central region of Chile. Because women are twice as likely to have gallstones and twice as likely to have gallbladder cancer as men, we plan to maximize our screening efficiency and number of outcomes by screening and enrolling women only. This approach is reasonable given that the female gender bias for gallbladder cancer is largely thought to be due to the gender bias for gallstones,1-3 suggesting that in the presence of gallstones, the risk of gallbladder cancer is the same for men and women. In addition, Chile is conducting a general population cohort in a small town in the high-risk area, and we can use the men with gallstones enrolled by the Chilean study to compare to the women in our study. We plan to enroll women with gallstones over 2 years and follow them for 6 years, conducting visits every other year to collect data on the primary exposures of interest, inflammatory markers and ultrasound characteristics, as well as additional exposures of interest, such as infections, genetics, and environmental exposures (e.g., aflatoxin, pesticides).

ELIGIBILITY:
* INCLUSION CRITERIA:

General Population Cohort:

* Female
* Age 50 years to 74 years
* No previous cholecystectomy
* Covered by National Health Insurance
* Resident of Araucania (or Maule)
* Able to answer questionnaire (due to language/communication issues or mental incapacity)

Other control (general population or cholecystectomy):

* No previous cholecystectomy
* Covered by National Health Insurance
* Resident of Araucania (or Maule)
* Able to answer questionnaire (due to language/communication issues or mental incapacity)

Gallbladder Cancer Group:

* Diagnosis within study time period
* Primary site of cancer is the gallbladder with histological or radiological confirmation
* Covered by National Health Insurance
* Resident of Araucania (or Maule)
* Able to answer questionnaire (due to language/communication issues or mental incapacity)

EXCLUSION CRITERIA:

General Population Cohort:

* Male
* Age less than 50 years or greater than 74 years
* History of previous cholecystectomy
* Not covered by National Health Insurance
* Not a Resident of Araucania (or Maule)
* Unable to answer questionnaire (due to language/communication issues or mental incapacity)

Other control (general population or cholecystectomy):

* History of previous cholecystectomy
* Not covered by National Health Insurance
* Not a Resident of Araucania (or Maule)
* Unable to answer questionnaire (due to language/communication issues or mental incapacity)

Gallbladder Cancer Group:

* Diagnosis not within study time period
* Primary site of cancer is NOT the gallbladder with histological or radiological confirmation
* Not covered by National Health Insurance
* Not a Resident of Araucania (or Maule)
* Unable to answer questionnaire (due to language/communication issues or mental incapacity)

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subject identification will begin with a census of the target neighborhoods in Chile in the study areas. Potential participants will be contacted by study staff (healthcare assistants), who will conduct home visits. If participant is eligible, study staff will invite the individual to participate and obtain written informed consent. She will then schedule an appointment at the study center for the screening ultrasound and give her the instructions to prepare for the examination.
Sampling Method: Non-Probability Sample
Enrollment: 4749 (Estimated)
Dates: Start 2017-01-11 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Cancer/precancer | during course of the study
  Our major exposures of interest are patterns, levels, and changes in inflammatory markers and ultrasound characteristics, with Gallbladder Dysplasia and Cancer as the primary outcome of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Jill E. Koshiol, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- Chile (3):
  - Hospital Regional de Talca, Talca
  - Universidad Catolica del Maule, Talca
  - Hospital Regional de Temuco, Temuco